CLINICAL TRIAL: NCT02118532
Title: The IN.PACT SFA Clinical Study for the Treatment of Atherosclerotic Lesions in the Superficial Femoral Artery and/or Proximal Popliteal Artery Using the IN.PACT Admiral™ Drug-Eluting Balloon in a Chinese Patient Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN.PACT SFA China
Record Dates: First submitted 2014-04-11; First posted 2014-04-21 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis; Superficial Femoral Artery; Proximal Popliteal Artery
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IN.PACT Admiral (Experimental)
  Interventions: Device: IN.PACT Admiral Paclitaxel-Eluting Percutaneous Transluminal Angioplasty (PTA) Balloon Catheter

INTERVENTIONS:
Device: IN.PACT Admiral Paclitaxel-Eluting Percutaneous Transluminal Angioplasty (PTA) Balloon Catheter — IN.PACT Admiral Paclitaxel-Eluting Percutaneous Transluminal Angioplasty (PTA) Balloon Catheter originally developed, approved and commercialized by Invatec Technology Center GmbH is the investigational medical device used in the study. Medtronic Inc. acquired Invatec on April 21, 2010. Medtronic

SUMMARY:
The purpose of this study is to confirm that the IN.PACT Admiral is safe and effective for the interventional treatment of new and non-stented restenotic lesions in the superficial femoral artery (SFA) and proximal popliteal artery (PPA) in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 85 years.
* Subject with documented diagnosis of peripheral arterial disease (PAD) classified as Rutherford class 2-3-4 in the superficial femoral artery (SFA) and/or proximal popliteal artery (PPA) above the knee, located in the arterial segment starting at least 1 cm beyond the Common femoral artery (CFA) bifurcation between the superficial and profunda femoris arteries (proximal anatomical landmark to the distal P1 segment of the popliteal artery at the level of the proximal edge of the patella (distal anatomical landmark).
* Target lesion consists of a single de novo or non-stented restenotic lesion (or a tandem lesion) or is a combination lesion
* Reference vessel diameter ≥ 4 mm and ≤ 7 mm by visual estimate.
* Subject able to walk without assistive devices (e.g. walker, cane).
* If subject has ipsilateral/contralateral iliac disease that requires treatment during the index procedure
* Angiographic evidence of adequate distal run-off to the foot (at least one native calf vessel [posterior tibial, anterior tibial, or peroneal arteries] is patent, defined as < 50% diameter stenosis).
* Female subjects of childbearing potential must have a negative pregnancy test ≤ 7 days before index procedure and willing to use a reliable method of birth control for the duration of the study or must have documented adequate birth control.
* Signed and dated Patient Informed Consent (PIC) form.
* Understands and accepts the duration of the study and is able and willing to comply with all requirements, including follow-up visits and evaluations.
* Life expectancy, in the Investigator's opinion, of at least 12 months.

Exclusion Criteria:

* In the investigator's opinion subject is unlikely to comply with the followup schedule.
* Stroke or STEMI within the 3 months prior to index procedure.
* Either local or systemic thrombolytic therapy within 48 hours prior to the index procedure.
* Inability to tolerate oral anticoagulation therapy (blood thinners such as warfarin) while on concomitant dual antiplatelet therapy (DAPT).
* Known allergies or sensitivities to heparin, aspirin (ASA), other anticoagulant/anti-platelet therapies, and/or paclitaxel or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.
* Breastfeeding woman.
* Chronic renal insufficiency with serum creatinine > 2.5 mg/dL within 14 days prior to index procedure.
* WBC < 3.0 (3,000 cells/mm3) within 14 days prior to index procedure.
* PLT count < 80,000 cells/mm3 or > 700,000 cells/mm3 within 14 days prior to index procedure.
* Known or suspected active systemic infection evidenced by WBC > 14.0 (14000/mm3) within 14 days prior to index procedure.
* Diagnosed with bleeding diatheses or hypercoagulable state.
* Subject is enrolled in another investigational device, drug or biologic study or subject was previously enrolled to the IN.PACT SFA China trial.
* Any major (e.g., cardiac. peripheral, abdominal) surgical procedure or intervention performed within 30 days prior to the index procedure.
* Any major (e.g., cardiac. peripheral, abdominal) elective procedure or intervention within 30 days post index procedure.
* Contralateral SFA/PPA disease requiring treatment in the same setting as index procedure.
* Presence of additional lesions in the target vessel that require treatment during index procedure but do not meet the definitions of tandem lesions.
* Target lesion is an in-stent or post-DEB restenosis or has been previously treated with bypass surgery.
* Failure to successfully cross the target lesion with a guide wire
* Lesion within or adjacent to an aneurysm.
* Acute or sub-acute thrombus in the target vessel.
* Angiographic evidence of severe calcification
* Target lesion known in advance of enrollment to require treatment with alternative therapy such as drug-eluting stent (DES), drug-eluting balloon (DEB), laser, atherectomy, cryoplasty, re-entry devices, cutting/scoring balloon, brachytherapy. Use of embolic protection devices is also prohibited.
* Pre-dilation resulted in a major ( ≥ Grade D) flow-limiting dissection (observed on 2 orthogonal views) or residual stenosis > 70% and translesional peak gradient > 10mm Hg.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Primary effectiveness endpoint: Primary patency within 12 months post-index procedure | 12 months
  Primary patency is defined as freedom from clinically-driven target lesion revascularization (TLR)1 and freedom from restenosis as determined by duplex ultrasound (DUS) Peak Systolic Velocity Ratio (PSVR) ≤ 2.4
Primary Safety Endpoint | 30 days post-index procedure
  A composite of freedom from device- and procedure-related mortality, freedom from major target limb amputation and freedom from clinicallydriven TLR within 30-day post-index procedure

SECONDARY OUTCOMES:
Major Adverse Events | 12 months
  MAE is defined as all-cause mortality, clinically-driven Target Vessel Revascularization (TVR), major target limb amputation or thrombosis at the target lesion site, through 12 months
Death of any cause | 30 days, 6 and 12 months
  Death of any cause at 30 days, 6 and 12 months
Target Lesion Revascularization | 30 days, 6 and 12 months
  Clinically-driven TLR at 30 days, 6 and 12 months TLR at 6 and 12 months
Target Vessel Revascularization | 30 days, 6 and 12 months
  Clinically-driven TVR at 30 days, 6 and 12 months TVR at 6 and 12 months
Major target limb amputation | 30 days, 6 and 12 months
  Major target limb amputation at 30 days, 6 and 12 months
Thrombosis at the target lesion site | 30 days, 6 and 12 months
  Thrombosis at the target lesion site at 30 days, 6 and 12 months
Time to first clinically-driven Target Lesion Revascularization | 12 months
  Time to first clinically-driven TLR through 12 months post-index procedure
Primary sustained clinical improvement | 6 and 12 months
  Primary sustained clinical improvement is defined as sustained upward shift of at least 1 category on Rutherford classification as compared to baseline without the need for repeated TLR or surgical revascularization in amputation-free surviving subjects.
Secondary sustained clinical improvement | 6 and 12 months
  Secondary sustained clinical improvement is defined as sustained upward shift of at least 1 category on Rutherford classification as compared to baseline including the need for repeated TLR or surgical revascularization in amputation-free surviving subjects.
Duplex-defined binary restenosis (PSVR > 2.4) of the target lesion | 6 and 12 months
  Duplex-defined binary restenosis (PSVR > 2.4) of the target lesion at 6 and 12 months post-index procedure, or at the time of reintervention prior to any pre-specified time point
Duplex-defined binary restenosis (PSVR > 3.4) of the target lesion | 6 and 12 months
  Duplex-defined binary restenosis (PSVR > 3.4) of the target lesion at 6 and 12 months post-index procedure, or at the time of reintervention prior to any pre-specified time point
Walking capacity assessment | 30 days, 6 and 12 months
  Walking capacity assessment by Walking Impairment Questionnaire (WIQ) at 30 days, 6 and 12 months
Walking distance | 30 days, 6 and 12 months
  Walking distance as assessed by 6 Minute Walk Test (6MWT) at 30 days, 6 and 12 months as change from baseline
Quality of life assessment | 30 days, 6 and 12 months
  Quality of life assessment by EQ5D questionnaire at 30 days, 6 and 12 months as change from baseline
Device success | Post procedure
  Device success is defined as successful delivery, balloon inflation, deflation and retrieval of the intact study device without burst below the rated burst pressure (RBP).
Procedural success | Post procedure
  Procedural success is defined as residual stenosis of ≤ 50% (non-stented subjects) or ≤ 30% (stented subjects) by core lab assessment.
Clinical success | Post procedure
  Clinical success is defined as procedural success without procedural complications (death, major target limb amputation, thrombosis of the target lesion, or TVR) prior to discharge.
Days of hospitalization due to the target lesion | 6 and 12 months
  Days of hospitalization due to the target lesion from procedure through 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Chen, Prof, Principal Investigator — Vascular Department Anzhen Hospital, Capital Medical University; Wei Guo, Prof, Principal Investigator — Vascular Department 301 Hospital
Locations (15):
- China (15):
  - 301 Hospital/Chinese PLA General Hospital, Beijing
  - Anzhen Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - West China Hospital, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Affiliated Hospital, Dalian Medical University, Dalian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The 1stAffiliated Hospital of Sun Yat-sen University, Guangzhou
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin
  - The first affiliated Hospital of Harbin Medical University, Harbin
  - Nanjing Drum Tower Hospital, Nanjing
  - Shanghai 9th People Hospital Affiliated Shanghai Jiao Tong University School of Medecine, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang

REFERENCES:
- [Derived] Shishehbor MH, Schneider PA, Zeller T, Razavi MK, Laird JR, Wang H, Tieche C, Parikh SA, Iida O, Jaff MR. Total IN.PACT drug-coated balloon initiative reporting pooled imaging and propensity-matched cohorts. J Vasc Surg. 2019 Oct;70(4):1177-1191.e9. doi: 10.1016/j.jvs.2019.02.030. PMID 31543165
- [Derived] Chen Z, Guo W, Jiang W, Wang F, Fu W, Zou Y, Deckers S, Li P, Popma JJ, Jaff MR. IN.PACT SFA Clinical Study Using the IN.PACT Admiral Drug-Coated Balloon in a Chinese Patient Population. J Endovasc Ther. 2019 Aug;26(4):471-478. doi: 10.1177/1526602819852084. Epub 2019 Jun 17. PMID 31204595
- [Derived] Schneider PA, Laird JR, Doros G, Gao Q, Ansel G, Brodmann M, Micari A, Shishehbor MH, Tepe G, Zeller T. Mortality Not Correlated With Paclitaxel Exposure: An Independent Patient-Level Meta-Analysis of a Drug-Coated Balloon. J Am Coll Cardiol. 2019 May 28;73(20):2550-2563. doi: 10.1016/j.jacc.2019.01.013. Epub 2019 Jan 25. PMID 30690141